CLINICAL TRIAL: NCT02555176
Title: A Pilot Trial of a Low-Carbohydrate Normocaloric Diet, in Patients With Head and Neck Carcinoma (HNC) and Its Effect on Stromal-Epithelial Metabolic Uncoupling
Brief Title: Low-Carbohydrate Normocaloric Diet in Patients With Head and Neck Carcinoma (HNC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15D.365; JT 5741 (Other: JeffTrial Number)
Record Dates: First submitted 2015-09-09; First posted 2015-09-21 (Estimated); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Carcinoma
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low Carbohydrate Diet (Experimental): Patients follow a normocaloric, low-carbohydrate diet for 10-28 days (from the time of cancer diagnosis to definitive surgical treatment).
  Interventions: Dietary Supplement: Dietary intervention

INTERVENTIONS:
Dietary Supplement: Dietary intervention — Follow a low-carbohydrate diet

SUMMARY:
This pilot clinical trial studies the effects of a low carbohydrate diet on tumor metabolism in patients with head and neck cancer. A low carbohydrate diet may reduce the metabolic activity of cancer cells and of surrounding supportive tissues. Studying samples of tissue and blood from patients with head and neck cancer in the laboratory before and after a low carbohydrate diet may help determine any changes in tumor metabolism.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the impact of a low-carbohydrate normocaloric diet on transporter of the outer mitochondrial membrane subunit 20 (TOMM20) expression by immunohistochemistry (IHC) in carcinoma cells and the impact of a low-carbohydrate normocaloric diet on monocarboxylate transporter 4 (MCT4) expression in fibroblasts.

SECONDARY OBJECTIVES:

I. Assess the feasibility of a low-carbohydrate normocaloric diet treatment in head and neck carcinoma (HNC) patients.

II. Assess the effect of a low-carbohydrate normocaloric diet on the serum levels of insulin, and insulin growth factor (IGF)-1 and -2.

III. Assess the potential impact of a low-carbohydrate normocaloric diet on the following: disease-free survival, distant metastases-free survival, overall survival.

IV. To evaluate the utility of cancer-derived exosomes to serve as prognostic biomarkers for real-time monitoring of therapeutic efficacy and identifying early recurrence using longitudinal samples from cancer patients undergoing treatment.

OUTLINE:

Patients follow a normocaloric, low-carbohydrate diet for 10-28 days (from the time of cancer diagnosis to definitive surgical treatment).

After completion of study, patients are followed up at 1 month, 3 months, and then every 3 months for 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of head and neck cancer biopsy proven, and who have a scheduled appointment for definitive resection of the tumor at TJUH are eligible to participate.
2. Subjects must be ≥ 18 and ≤ 70 years of age.
3. KPS > 70
4. Expected survival > 6 months.
5. Adequate organ functions (hematological, hepatic, renal function).
6. Absolute neutrophil count > 1.5 x 109/L, platelet count > 100 x 109/L, hemoglobin > 9 g/L, total bilirubin < 1.25 x the institutional upper limit of normal [ULN], albumin > 2.5 g/dL, aspartate aminotransferase < 45 IU/dL, alanine aminotransferase < 40 IU/dL, alkaline phosphatase ≤ 190 IU/dL and serum creatinine < 1.3 mg/dL and creatinine clearance > 50 mL/min.
7. Serum potassium and magnesium, and corrected serum calcium within the institution's normal reference range.
8. Ability to provide written informed consent obtained prior to participation in the study.
9. Women of childbearing potential (WOCBP) must be willing to use an adequate method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized.
10. Patients' availability to check their weight twice per week, during the study duration.

Exclusion Criteria:

1. Diabetic patients are eligible but will be excluded if they are taking metformin, insulin or sulfonilureas.
2. Patients with plasma alanine aminotransferase greater than 40 IU/dL.
3. Patients with plasma aspartate aminotransferase greater than 45 IU/dL.
4. Patients with plasma creatinine level greater than 1.3 mg/dL.
5. Patients with plasma alkaline phosphatase greater than 190 IU/dL.
6. Patients with plasma bicarbonate less than 22 mEq/L or history of lactic or any other metabolic acidosis.
7. Patients with history of congestive heart failure.
8. Patients with myocardial ischemia or peripheral muscle ischemia.
9. Patients with sepsis or severe infection.
10. Patients with history of lung disease currently requiring any pharmacologic or supplemental oxygen treatment.
11. Patients scheduled for definitive HNC cancer surgical resection less than 10 days from enrollment or greater than five weeks from enrollment.
12. Patients with history of hepatic dysfunction or hepatic disease.
13. Patients with a history of excessive alcohol intake which is defined in accordance with CDC definitions as more than 1 drink per day for women and more than 2 drinks per day for men. This definition is referring to the amount consumed on any single day and is not intended as an average over several days. A standard drink is equal to 13.7 grams (0.6 ounces) of pure alcohol. Generally, this amount of pure alcohol is found in 12-ounces of beer, 8-ounces of malt liquor, 5-ounces of wine, 1.5-ounces or a "shot" of 80-proof distilled spirits or liquor (e.g., gin, rum, vodka, or whiskey).
14. Patients with a lower BMI (BMI<18) will be excluded.
15. Patients with history of known defects in fat metabolism (ie pyruvate carboxylase deficiency, prophyria, fatty acid oxidation defects, primary carnitine deficiencies, organic acidurias, hypoglicemia) will be excluded.
16. Pregnancy, lactation or inability to use medically acceptable birth control if of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change in TOMM20 expression by IHC | Baseline to up to 28 days (day of surgery)
  IHC status will be classified as positive or negative pre-and post-treatment. Change in IHC status will be evaluated using McNemar's test for paired dichotomous data.
Change in MCT4 expression in fibroblasts | Baseline to up to 28 days (day of surgery)
  IHC status will be classified as positive or negative pre-and post-treatment. Change in IHC status will be evaluated using McNemar's test for paired dichotomous data.
Incidence of adverse events, evaluated using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0 | Up to 24 months after surgery

SECONDARY OUTCOMES:
Feasibility of a low-carbohydrate normocaloric diet treatment in HNC patients | Up to 28 days
  Analysis will be descriptive
Change in serum levels of insulin | Baseline to up to 24 months
Change in serum levels of IGF-1 | Baseline to up to 24 months
Change in serum levels of IGF-2 | Baseline to up to 24 months
Disease-free survival | Up to 24 months after surgery
  Estimated using the Kaplan-Meier method.
Distant metastases-free survival | Up to 24 months after surgery
  Estimated using the Kaplan-Meier method.
Overall survival | Up to 24 months after surgery
  Estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Curry, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Jefferson University Hospitals — http://hospitals.jefferson.edu/